CLINICAL TRIAL: NCT06704126
Title: A Crossover Study of Passive Movement Training, With and Without Blood Flow Restriction, to Examine Postprandial Blood Glucose Levels
Brief Title: Does Passive Movement Increase Glucose Uptake Into Muscle?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lancaster University (Other)
Responsible Party: Principal Investigator, Paul Hendrickse, Lecturer in Biomedicine, Lancaster University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: FHM-2024-4434-SA-2
Record Dates: First submitted 2024-11-19; First posted 2024-11-25 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Glucose; Insulin; Blood Flow Restriction Therapy; Blood Flow Velocity
Keywords: Passive movement training; Blood flow restriction; Glucose; Insulin; Passive movement
MeSH Terms: conditions — Insulin Resistance | interventions — Range of Motion, Articular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Passive movement only (Experimental): Participants undergo passive movement training only
  Interventions: Other: Passive movement
- Passive movement + intermittent blood flow restriction (Experimental): Participants undergo passive movement training with blood flow restriction applied intermittently during the passive movement protocol
  Interventions: Other: Passive movement with blood flow restriction
- Control (No Intervention): Sitting still in Biodex only - no movement

INTERVENTIONS:
Other: Passive movement — This study will use a passive movement protocol delivered on a Biodex isokinetic dynamometer at 1Hz for 60 seconds on, 60 seconds off, for a total of 30 minutes.
  Arms: Passive movement only
Other: Passive movement with blood flow restriction — This study will use a passive movement protocol delivered on a Biodex isokinetic dynamometer at 1Hz for 60 seconds on, 60 seconds off, for a total of 30 minutes. During the 60 seconds on of passive movement training, blood flow restriction cuffs which will be applied to the legs, will be inflated to cause 80% arterial blood flow occlusion.
  Arms: Passive movement + intermittent blood flow restriction

SUMMARY:
This study aims to examine the blood sugar response after a meal, and how three different movement protocols may impact the blood sugar level.

Participants will visit the lab on three different occasions. Before each visit the participant will eat a meal we give them and have a cannula (a needle with a tube) put in their arm to allow blood sampling for the visit.

Visit A will be the participant just having their legs moved by the machine, visit B will be the participant having their legs moved by the machine with the addition of blood pressure cuffs on their thighs, and visit C will just be the participant sitting still on the machine.

DETAILED DESCRIPTION:
This study will require nine participants to be recruited and enrolled. The aim of the study is to determine the effect of passive movement, with and without blood flow restriction, on blood glucose and insulin primarily. Other outcomes included elsewhere in this registration. The protocol will involve an initial health screening/familiarisation session in the Human Performance Laboratory (HPL) at Lancaster University, followed by three randomly ordered HPL visits per participant. At the beginning of each HPL visit, the participant will be given a standard meal. The design is a crossover study therefore each participant will complete visits A, B and C and act as their own control.

Each of the visits A, B and C will involve consumption of a meal (86g carbohydrate content) and insertion of a cannula to the arm. Blood samples will then be drawn from the cannula at five minute intervals for approximately 3.5 hours. Three gold-top vacutainers will be taken throughout each visit to allow for insulin analysis. Once the blood is sampled, the vacutainer will be left to clot at room temperature for 15 minutes and then spun in a centrifuge at 4°C, 1800 RCF, for 10 minutes. The supernatant will be transferred to a microfuge tube via pipetting and stored at -80°C until analysis at a future date using an enzyme-linked immunosorbent assay (ELISA). In addition, 1ml syringe blood samples will be taken every 5 minutes and ejected onto a non-absorbent pad. A fraction of this ejection on the pad will then drawn up into a capillary tube to be analysed by a Biosen benchtop glucose/lactate analyser.

Visit A will invole the participant sitting on a Biodex isokinetic dynamometer and having both legs passively flexed and extended through 90 degrees, at a frequency of 1Hz for 30 minutes. This will be 60 seconds on, followed by 60 seconds off, repeated 15 times.

Visit B will involve the same as visit A, but with the addition of blood flow restriction intermittently. These are blood pressure bands (VALD AirBands) around the thighs which will inflate and deflate to cause 80% arterial occlusion in their inflated state. These will inflate and deflate in tandem with the passive movement going on and off.

Visit C is a control visit and will involve the participant sitting in the Biodex only with no movement or blood flow restriction occuring.

Throughout the study, measurements will be taken to meausure the outcome measure specified in this registration.

ELIGIBILITY:
Inclusion Criteria:

* 18-35 years old, inclusive
* Male
* Healthy (no known long-term health conditions / acute febrile illness)

Exclusion Criteria:

* Smokers
* Recent blood donation (within 12 weeks)
* Any medication
* Phobia of needles
* Blood pressure ≥ 140/90 mmHg, either figure
* Any potential atrial fibrillation or cardiovascular health conditions
* Diabetes
* Allergies to barley, gluten, nuts, almonds

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-07-11 (Actual); Study Completion 2025-07-11 (Actual)

PRIMARY OUTCOMES:
Blood glucose level | From pre-meal, every 5 minutes for 150 minutes
  Obtained by 5 minute interval blood draws from cannula then drawn up by a capillary tube and analysed by Biosen benchtop analyser

SECONDARY OUTCOMES:
Blood insulin level | Immediately pre-meal, 30 minutes post-meal and 60 minutes post-meal
  Obtained by gold-top vacutainer blood draw
Blood lactate level | From pre-meal, every 5 minutes for 150 minutes
  Obtained by 5 minute interval blood draws from cannula then drawn up by a capillary tube and analysed by Biosen benchtop analyser
Femoral arterial blood velocity | Measured at 0, 1, 5, 10, 20 and 30 minutes relative to the movement/control protocol commencing
  Obtained pulse speed via ultrasound doppler
Electromyography | Measured for 30 minutes beginning from movement/control protocol commencement
  Electromyography used to obtain magnitude of voluntary muscle contraction, sensor placed at 80% on the line between the anterior spina iliaca superior and the joint space in front of the anterior border of the medial ligament with perpendicular orientation as per Seniam guidance

OTHER OUTCOMES:
Muscular thickness | Measured immediately post-meal and then again 30 minutes post-meal, on each of the three visits.
  Muscle thickness of the quadriceps femoris to be measured using a B-mode ultrasonography with a linear-array probe. Muscle thickness to be determined as the distance between the muscle fasciae and bone interface, and the sum of measurements of the 8 sites used in the analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Hendrickse, PhD, Principal Investigator — Lancaster University
Locations (1):
- Lancaster University, Lancaster, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No benefit to sharing these data.